CLINICAL TRIAL: NCT02941666
Title: Human Mesenchymal Stem Cells in the Synovial Fluid of the Hip in Patients With Osteonecrosis of the Femoral Head
Brief Title: Human Mesenchymal Stem Cells in the Synovial Fluid of the Hip
Status: Terminated | Type: Observational
Why Stopped: Study staff was unable to collect proper samples to meet study goals
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rafael J. Sierra, M.D., Professor of Orthopedics, Mayo Clinic
Other Study IDs: 16-002241
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Osteonecrosis
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Collapse ON group: This group will consist of patients who have concentrations of Mesenchymal Stem Cells in with post collapse osteonecrosis.
- Pre-collapse group: This group will consist of patients who have concentrations of Mesenchymal Stem Cells in with pre-collapse osteonecrosis.
- FAI group: This control group will be selected in patients undergoing hip arthroscopy for femoral/acetabular impingement.

SUMMARY:
Previous studies have shown an increase in the concentration of mesenchymal stem cells (MSC's) in the setting of osteoarthritis of the knee and its correlation to severity. Researchers have shown that as there is an increase in the severity of the disease, the concentration of stem cells also increases. The purpose of this study is to determine if there is the same increase in stem cell concentration in patients with osteonecrosis (ON) of the femoral head.

DETAILED DESCRIPTION:
Since the treatment of osteonecrosis is related to the severity of disease, namely articular cartilage collapse, the purpose of this study is to determine if the MSC concentration in synovial fluid can be correlated to disease stage. In order to do this the investigators will:

Milestone #1:

Determine the concentration of MSC's in the synovial fluid in patients with osteonecrosis. This work will be carried out utilizing FACS-based technique to synovial fluid stem cell sub-population.

Milestone #2:

Compare concentrations of MSC's in patients with pre collapse, post collapse osteonecrosis and "normal" hips. Patient-derived MSC will be quantified at the different stages of disease and assays will be performed in order to assess their viability. A control group will be selected in patients undergoing hip arthroscopy for femoral/acetabular impingement (FAI). Since FAI does not affect the intraarticular environment of the hip, theoretically these patients would have a "normal" concentration of synovial stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients consented to undergo a THA (post-collapse osteonecrosis), hip arthroscopy or minimally invasive core decompression
* Preoperative radiographic diagnosis of ON or FAI (femoral/acetabular impingement)

Exclusion Criteria:

* Pregnant females
* Active infection, HIV, Hepatitis C or B, syphilis Immunodeficiency
* Patients receiving hematopoetic growth factors or anti-angiogenesis products

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in clinic as scheduled for total hip arthroplasty, hip arthroscopy or minimally invasive core decompression of the femoral head after granting consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
The quantity of mesenchymal stem cells present in the synovial fluid of patients with precollapse ON of the femoral head and postcollapse ON of the femoral head compared to patients without intraarticular hip pathology. | 24 months
  Previous studies have shown an increase in the concentration of MSCs in the setting of osteoarthritis of the knee and its correlation to severity. Researchers have shown that as there is an increase in the severity of the disease, the concentration of stem cells also increases. The purpose of this study is to determine if there is the same increase in stem cell concentration in patients with osteonecrosis (ON) of the femoral head. Since the treatment of osteonecrosis is related to the severity of disease, namely articular cartilage collapse, the purpose of this study is to determine if the MSC concentration in synovial fluid can be correlated to disease stage.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael J. Sierra, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials